CLINICAL TRIAL: NCT05278247
Title: An Open Single-center Study in England to Assess Safety and Performance of a NIRS System to Monitor Abdominal Tissue Oxygen Saturation in Preterm Infants
Brief Title: Sensing Oxygen Saturations Using Abdominal NIRS With an Investigational Realtime Device (Songbird)
Acronym: (Songbird)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carag AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021.9635
Record Dates: First submitted 2022-02-22; First posted 2022-03-14 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: NEC
Keywords: abdominal NIRS for oxygen saturation

STUDY DESIGN:
Intervention Model Description: confirmatory, open, single-arm, mono-centric
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm for all subjects (Experimental): all subjects receive the same diagnostic measurement
  Interventions: Diagnostic Test: NIRS

INTERVENTIONS:
Diagnostic Test: NIRS — Performance of a NIRS to monitor abdominal tissue oxygen saturation in preterm infants

SUMMARY:
Preterm infants are highly vulnerable and may suffer from multiple life-threatening conditions that manifest low tissue oxygenation (StO2). Near infrared spectroscopy (NIRS) is a technique available to non-invasively and safely monitor the tissue oxygenation status (StO2), which can be beneficial or live saving for this fragile patient population. Unfortunately, traditional NIRS devices show a broad variability when applied to the abdomen (Bailey & Mally 2016). The novel device is designed especially for application of NIRS on the abdomen of preterm infants.

DETAILED DESCRIPTION:
Each child will be measured over a time span of three days with the novel NIRS device.

1. A two-hour measurement is performed in measurement phase 1
2. Additionally, the sensor will be placed five times onto the abdomen for 1-minute measurements, which constitutes measurement phase 2.
3. The final measurement phase 3 lasts for up to 70 hours.

A total of two ultrasound (US) examination on the abdomen are performed during the first two measurement phases to assess the presence of air and stool in the abdomen.

Additional assessment of SpO2 is performed throughout. Aside from the US and SpO2 measurement, no additional procedures will be performed.

The NIRS measurement will not disturb necessary clinical and nursing procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infants with Gestational age less than 35 0/7 weeks
2. Signed Informed consent of the legal representative(s) is received after being informed. The consent form is signed by one legal representative, which is likely to be either the mother or the father. Only married fathers or those listed on the birth certificate are considered under UK regulations. In the case of non-married father, the mother must provide consent.
3. Clinically stable condition. The clinical stability is to be reconfirmed before the start and checked during the measurement.

Exclusion Criteria:

1. Injured, hypersensitive or bruised skin present on the abdomen,
2. Existence of clinical instability at any time during the investigation leads to exclusion, if ordered so by the physician entrusted with the investigation,
3. Any medical care equipment, e.g. patches, dressing, umbilical arterial or venous catheter, blood supply, etc., prohibiting correct placement of the sensors,
4. Severe Congenital malformations,
5. Clinical abdominal concerns
6. Severe metabolic disorders,
7. Early onset sepsis,
8. Inability of legal representatives to understand the purpose of the clinical trial due to language barriers such as the insufficient ability to understand the spoken or written language,
9. The treatment of newborn jaundice with light during measurement time phase 1 and 2,
10. Previous enrolment into the current study,
11. Family members, employees and other dependent persons of the investigator,
12. Participation in another study with investigational drug/device within the preceding days and during the present study which may influence abdominal oxygen saturation.
13. Known silicone allergy

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Performance of the CTOM system | 3 days
  We intend to investigate sensor handling on preterm infants and record the signal variability and reproducibility. A measurement signal serves to analyse reproducibility, signal quality and different signal analysis methods.
  Abdominal oxygen tissue saturation will be calculated. The aStO2 values will be calculated with and without considering the presence of additional absorbers besides haemoglobin. The datasets to be analysed include three measurement series per subject from a total of at least 50 subjects. The planned analyses consist of descriptive statistics and time series analysis.

SECONDARY OUTCOMES:
Occurrence of adverse events is measured | 3 days
  AEs will be recorded and analyzed with regards to their relationship to the investigational device and the measurement procedure. The occurrence of adverse events, especially skin markers, will be measured. The study will compare AEs and SAEs from this study with documented AEs and SAEs employing NIRS devices.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Chapman, Study Chair — lead NHS R&D contact

IPD SHARING:
Plan to Share IPD: No